CLINICAL TRIAL: NCT02882256
Title: Video Discharge Instructions (VDI) as Adjuncts to Written Discharge Instructions for 3 Common Chief Complaints in the Emergency Department (ED)
Brief Title: Video Discharge Instructions (VDI) as Adjuncts to Written Discharge Instructions in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Melissa McCarthy, Associate Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 061612
Record Dates: First submitted 2016-08-04; First posted 2016-08-29 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Urinary Tract Infection; Head Injury; Laceration
Keywords: laceration; urinary tract infection; minor head injury; concussion
MeSH Terms: conditions — Urinary Tract Infections; Craniocerebral Trauma; Lacerations; Brain Concussion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients will receive video discharge instructions in addition to standard written discharge instructions.
  Interventions: Other: Video discharge instructions
- Control (No Intervention): Patients will receive standard written discharge instructions.

INTERVENTIONS:
Other: Video discharge instructions — Discharge instructions provided in video form
  Arms: Intervention

SUMMARY:
Patients seen in the ED with either a laceration, minor head injury, or urinary tract infection will be randomized to one of two groups. Both groups will receive the standard written discharge instructions; in addition, one group will watch video discharge instructions. Each patient will be asked to complete a short survey with questions related to the discharge instructions received in the ED, and will be called 5-7 days after the ED visit to ask questions about discharge instructions and the ED visit.

DETAILED DESCRIPTION:
Patients will be enrolled in the study at George Washington University Hospital's Emergency Department. Patients who consent will be randomly assigned to one of two groups; (1) standard Written Discharge Instructions from the nursing staff (2) standard Written Discharge Instructions from the nursing staff AND watching the Video Discharge Instructions on a tablet. Subjects will complete a survey after they have received their discharge instructions and before leaving the ER. Several (5-7) days after leaving the Emergency Department, subjects will receive a phone call from one of the investigators staff members asking 2-3 questions about their ED visit and how they treated the condition at home. The survey questions at discharge and at follow-up will pertain to how to care for the condition and will be based on the discharge instructions. The study is designed to determine if patients retain health information more accurately if they watch a video in addition to being given written information. A total sample size of 200 participants will be recruited. Enrollment for this study will begin June of 2016 and will continue until the investigators have enough participants. The data analyst will be blinded to treatment assignment when analyzing the data.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age
* Patient speaks English fluently
* Patient was diagnosed with Urinary Tract Infection, Laceration, or Minor Head Injury

Exclusion Criteria:

* Patient is presently a prisoner or in police custody
* Patient unable to understand consent
* Patient does not have a cell phone or house line
* Patient is blind or hearing impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Understanding of discharge diagnosis using questionnaire | Immediately before leaving the emergency department for discharge home.
  Right after the provider who discharges the patient goes over the discharge instructions with the subject, the investigators will administer the discharge questionnaire.

SECONDARY OUTCOMES:
Patient satisfaction of overall care in ED using questionnaire | Five to seven days after the index ED visit.
  Subjects will complete a telephone follow-up interview 5-7 days after ED discharge.
Self-reported compliance with post-discharge care using questionnaire | Five to seven days after the index ED visit.
  Subjects will complete a telephone follow-up interview 5-7 days after ED discharge.
Comprehension of return precautions using questionnaire | Five to seven days after the index ED visit.
  Subjects will complete a telephone follow-up interview 5-7 days after ED discharge.
Retention of understanding of discharge diagnosis using questionnaire | Five to seven days after the index ED visit.
  Subjects will complete a telephone follow-up interview 5-7 days after ED discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Griffin Davis, MD, Principal Investigator — GW Medical Faculty Associates
Locations (1):
- George Washington University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bloch SA, Bloch AJ. Using video discharge instructions as an adjunct to standard written instructions improved caregivers' understanding of their child's emergency department visit, plan, and follow-up: a randomized controlled trial. Pediatr Emerg Care. 2013 Jun;29(6):699-704. doi: 10.1097/PEC.0b013e3182955480. PMID 23714763
- [Result] Atzema CL, Austin PC, Wu L, Brzozowski M, Feldman MJ, McDonnell M, Mazurik L. Speak fast, use jargon, and don't repeat yourself: a randomized trial assessing the effectiveness of online videos to supplement emergency department discharge instructions. PLoS One. 2013 Nov 11;8(11):e77057. doi: 10.1371/journal.pone.0077057. eCollection 2013. PMID 24244272